CLINICAL TRIAL: NCT03391245
Title: Vitamin D Level and Risk of Infections in Cirrhotic Patients: Does it Have a Role?
Brief Title: Vitamin D Level and Risk of Infections in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr. Nahed A. Makhlouf, Assistant Professor, Assiut University
Other Study IDs: VDLARIACP
Record Dates: First submitted 2017-12-27; First posted 2018-01-05 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Vitamin D Deficiency; Infection; Liver Cirrhosis
MeSH Terms: conditions — Vitamin D Deficiency; Infections; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhotic patients with or without infection: We will include admitted patients with liver cirrhosis irrespective of the underlying etiology during 6 months in Al Rajhi Tertiary Liver Hospital, Assiut, Egypt. They will be divided into 2 Groups. Group I: Cirrhotic patients with evidence of infections at any site and Group II: Cirrhotic patients without evidence of infections.
  Diagnosis of infection will based on related clinical symptoms and signs with laboratory and radiological findings.
  Interventions: Diagnostic Test: 3- Serum 25-Hydroxy Vitamin D level will be measured by Competitive ELISA technique

INTERVENTIONS:
Diagnostic Test: 3- Serum 25-Hydroxy Vitamin D level will be measured by Competitive ELISA technique — Serum 25-Hydroxy Vitamin D level will be measured by Competitive ELISA technique using CALBIOTECH (A life science company) kit, Catalog No.: VD220B

SUMMARY:
It is widely known that vitamin D has an important role in calcium metabolism and bone mineralization. Its deficiency is related to rickets and osteomalacia in children and adults respectively. Vitamin D had a role in innate and acquired immunity. It increases innate defense and modulates lymphocytes activation, leading to a change toward a T2 helper response ).

The role of vitamin D deficiency on the risk of bacterial infection among patients in intensive care units has been reported. An observational studies in children reported an association between low 25-OH vitamin D level and infectious viral diseases .

The deranged metabolism of vitamin D in liver cirrhosis was first reported in the late '70s and was attributed mainly to impaired 25(OH)-vitamin D hydroxylation of the precursor vitamin D caused by impaired liver function. Low level of vitamin D was found independently to be associated with increased risk of bacterial infections in patients with liver cirrhosis.

The observed relationship between the lack of vitamin D and the increase risk of mortality in cirrhotic patients could be attributed to bacterial infections. Thus, the association of low vitamin D levels with liver insufficiency and infections supports the use of vitamin D as a prognostic marker in the population of cirrhosis.

Studies on the role of vitamin D as a risk factor for infections in patients with liver cirrhosis are not well studied in our locality(Upper Egypt).

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients with liver cirrhosis irrespective of the underlying etiology during 6 months in Al Rajhi Liver Hospital, Assiut, Egypt who accept to participate in the study

Exclusion Criteria:

* Patients with cholestatic liver disease, patients receiving antibiotics to treat their infection prior hospital admission and patients refusing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include admitted patients with liver cirrhosis irrespective of the underlying etiology during 6 months in Al Rajhi Tertiary Liver Hospital, Assiut, Egypt. They will be divided into 2 Groups. Group I: Cirrhotic patients with evidence of infections at any site and Group II: Cirrhotic patients without evidence of infections.
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-02-15 (Estimated)

PRIMARY OUTCOMES:
Vitamin D deficiency as a risk factor for infection in cirrhotic patients | 6 month
  Measurement of Vitamin D levels in cirrhotic with infection when compared with cirrhotic without infection and determination of Vitamin D level cut-off points for infection in cirrhotic patients

SECONDARY OUTCOMES:
Correlation of Vitamin D level with Liver Disease severity | 6 month
  Correlation of Vitamin D level with Child Pugh Grade
Correlation of vitamin D level with liver disease severity | 6 month
  Correlation of Vitamin D level with MELD score
Determination of independent predictor of infection in cirrhotics | 6 month
  Use of logistic regression analysis for risk factors for infection in cirrhotic patients

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Mahmoud, M.D, Study Director — Assiut Uiversity
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided